CLINICAL TRIAL: NCT06628856
Title: Ex Ante and Interim Evaluation of the Quality of Life of the Piloted Persons, and Cost-efficiency Analysis
Brief Title: Quality of Life of the Piloted Individuals and a Cost-efficiency Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ACP 2/2023
Record Dates: First submitted 2024-02-26; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-02

CONDITIONS: Terminal Illness
Keywords: Person-centred care; meaningful activities; direct care professional; occupational therapist
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HOSPITAL CHILE (Experimental): The study proposes a 3-time longitudinal design, with evaluations at baseline, 2.5 months, and 5 months, to measure the impact of an intervention on terminally ill patients and their families, focusing on health status, quality of life, and emotional well-being. (N=286)
  Interventions: Other: Quality of life
- HOSPITAL SPAIN (Experimental): The study proposes a 3-time longitudinal design, with evaluations at baseline, 2.5 months, and 5 months, to measure the impact of an intervention on terminally ill patients and their families, focusing on health status, quality of life, and emotional well-being. (N=286)
  Interventions: Other: Quality of life

INTERVENTIONS:
Other: Quality of life — The study proposes a 3-time longitudinal design, with evaluations at baseline, 2.5 months, and 5 months, to measure the impact of an intervention on terminally ill patients and their families, focusing on health status, quality of life, and emotional well-being.

SUMMARY:
The increasing life expectancy and global aging population necessitate changes in long-term gerontological services based on Person-Centred Care approaches. This study aims to improve Person-Centred Care in geriatric centers through meaningful activities and the role of occupational therapists and direct care professionals in developing these activities. A descriptive cross-sectional quasi-experimental design was proposed, with 10 participants.

DETAILED DESCRIPTION:
Background: Increasing life expectancy means that the ageing of populations globally is on the rise. It is therefore important to promote changes in long-term gerontological services based on Person-Centred Care approaches, in which meaningful occupation serves as a basis and is supported by appropriate professional support, such as the occupational therapist and the direct care professional.

Objective: The study aims to analyze the needs, quality of life, and coping strategies of terminally ill patients over five months, as well as burnout and dehumanization among caregivers and healthcare staff.

Methods: This study examines factors influencing the quality of life (QOL) of terminally ill patients and the burnout and dehumanization of caregivers and health professionals using a mixed methodology. The study proposes a 3-time longitudinal design, with evaluations at baseline, 2.5 months, and 5 months, to measure the impact of an intervention on terminally ill patients and their families, focusing on health status, quality of life, and emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* That the direct care worker has a degree as a nursing assistant, dependency care technician, geroculturist or certificate of professionalism.
* The worker must speak and understand Spanish.
* The residence must offer service during the day, in the morning or afternoon shift.
* Workers must have been with the department for more than 4 months.

Exclusion Criteria:

* Workers who work night shift only.
* Workers on rotating shifts in all departments of the residence.
* Workers absent at the time of the study due to temporary leave, vacations or other causes.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 166 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Qualitative analysis | 5 MONTHS
  structured interviews: The coding system for the qualitative information will be carried out using the Atlas-Ti content analysis program. Atlas-Ti allows exporting a matrix to SPSS format, as a quantitative data matrix composed of the set of ideas, identified by the code of each interview, the idea number and its corresponding code for affected person and family member. In this way, the frequencies of the different categories can be analyzed.
Multilevel analysis | 5 MONTHS
  daily records: Multilevel analyses will be performed by applying Mix Models with maximum likelihood (ML) estimation.
Student's t-tests | 5 MONTHS
  telematic records: Student's t-tests for independent samples and ANOVAs/ANCOVAs will be applied to analyze differences in the study variables (needs, QOL, coping strategies) according to sociodemographic (sex, age, educational level) and clinical variables (type of disease, type of treatment or dependency status).

CONTACTS AND LOCATIONS:
Locations (1):
- Olalla Saiz Vazquez, Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No